CLINICAL TRIAL: NCT04172077
Title: Association Of Self Efficacy Levels, Resiliency Levels and Attachment Styles of Adolescents With Type 1 Diabetes and Their Caregivers
Brief Title: Self Efficacy Levels, Attachment Style and Resiliency of Youth With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Vanita Pais, Registered Dietitian, The Hospital for Sick Children
Other Study IDs: 1000059604
Record Dates: First submitted 2018-03-09; First posted 2019-11-21 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Type1diabetes
Keywords: Self Efficacy; Resiliency; Attachment style and youth with type 1 diabetes

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will assess self-efficacy levels(SE) ,resiliency and attachment style of adolescent with type 1 diabetes and their caregivers.SE and attachment style of patients and parents will be compared with each other as well as correlated with diabetes management as assessed by A1C and self inventory scale.

ELIGIBILITY:
Inclusion Criteria:

* T1DM patients age 12 - 18 yrs from Sick Kids Diabetes Clinic and a primary caregiver
* T1DM > 1yr and able to communicate in English

Exclusion Criteria:

* Families who cannot communicate in English (read, write, speak)
* Diagnosed less than 1 year diabetes
* Transient form of Diabetes (such as medication induced diabetes)
* Exclude type 2 Diabetes and CFRD (cystic fibrosis related diabetes)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: T1DM patients aged 12 - 18 yrs from Sick Kids Diabetes Clinic and their primary caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Examine the effects of patients' attachment styles (secure, mixed and fearful) on their type one diabetes management represented by A1C level | 25 minutes
  The following tool will be used - Relationship Scale Questionnaire (RSQ): The 30-item RSQ is valid and reliable. 76 Re-test reliability of the RSQ ranged from 0.54 to 0.78 and correlation coefficients of RSQ and RQ ranged from 0.41 to 0.6191.
  Adolescent Relationship Scale Questionnaire (A-RSQ): Sümer & Güngör (1999) used the A-RSQ and report validity of 0.7-0.95 as well as an internal consistency of 0.82.

SECONDARY OUTCOMES:
a) Effect of attachment style on self efficacy level in patients. | 25 minutes
  The following tool will be used - Self-Efficacy of Diabetes Self-Management (SEDM): This is a 10-item questionnaire that is used to assess perceived self-efficacy to preform diabetes care behaviours. Respondents are asked to score responses on a 1-10 Likert scale in which '1= not at all sure' to '10= completely sure'.
a) Effect of attachment style on self efficacy level in parents. | 25 minutes
  The following tool will be used - Self-Efficacy of Diabetes Self-Management (SEDM): This is a 10-item questionnaire that is used to assess perceived self-efficacy to preform diabetes care behaviours. Respondents are asked to score responses on a 1-10 Likert scale in which '1= not at all sure' to '10= completely sure'.
b)Compare diabetes management self-efficacy and attachment style in patients. | 25 minutes
  To compare diabetes self-efficacy (SEDM) in patients and their parents, paired t-tests will be calculated. In addition, to compare attachment styles in patients and their parents, McNemar's test will be used. Paired t-tests and McNemar's tests effectively take into account the correlations between parent-adolescent measures from the same family.
b)Compare diabetes management self-efficacy and attachment style in parents | 25 minutes
  To compare diabetes self-efficacy (SEDM) in patients and their parents, paired t-tests will be calculated. In addition, to compare attachment styles in patients and their parents, McNemar's test will be used. Paired t-tests and McNemar's tests effectively take into account the correlations between parent-adolescent measures from the same family.

CONTACTS AND LOCATIONS:
Overall Officials: Vanita Pais, BSc,CDE, Principal Investigator — Sick Kids Hospital; Christabelle Almeida, MSc,CDE, Study Director — Sick Kids Hospital
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No